CLINICAL TRIAL: NCT01125891
Title: Phase I Dose Escalation Study of Gemcitabine and ON 01910.Na in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Dose Escalation Study of Gemcitabine and ON 01910.Na in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-09; NCT00822939 (obsolete NCT alias)
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Malignant Neoplasmas; Solid Tumors
Keywords: gemcitabine hydrochloride; Gemzar; ON 01910.Na
MeSH Terms: interventions — Gemcitabine; ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine and ON 01910.Na (Experimental)
  Interventions: Drug: gemcitabine; Drug: ON 01910.Na

INTERVENTIONS:
Drug: gemcitabine — The dose of gemcitabine will be fixed at 1000 mg/m2 i.v. as a 30 minutes infusion on days 1, 8, and 15 every 28 days.
  Other Names: Gemzar
Drug: ON 01910.Na — The starting dose of ON 01910.Na is 600 mg/m2 as a 2 hour intravenous (i.v.) infusion on days 1, 4, 8, 11, 15 and 18 of a 28-day course. The dose of ON 01910.Na will be escalated in increments in successive cohorts (dose level (DL) 1 = 600 mg/m2, DL 2 = 1200 mg/m2, DL 3 = 1800 mg/m2) of new patients.
  Other Names: rigosertib sodium

SUMMARY:
Treatment of cancer is often more effective when two or more drugs are used together. For example, when gemcitabine, an approved drug, and ON 01910.Na, a new investigational anti-cancer drug, are used together to treat cancer cells in laboratory animals, there is more inhibition of the growth of the cancer cells compared to either drug used by itself. These results offer promise that gemcitabine and ON 01910.Na could be used to treat cancer in patients. However, before studies that seek to find out if gemcitabine and ON 01910.Na is an effective combination in patients can be done, doctors must first know what is largest, safe dose of ON 01910.Na that can be used in combination with gemcitabine. This study is designed to answer that question.

DETAILED DESCRIPTION:
The order of infusion on Days 1, 8, and 15 will be gemcitabine first, immediately followed by ON 01910.Na. The dose of gemcitabine will be fixed at 1000 mg/m2 i.v. as a 30 minutes infusion on days 1, 8, and 15 every 28 days. The starting dose of ON 01910.Na is 600 mg/m2 as a 2 hour intravenous (i.v.) infusion on days 1, 4, 8, 11, 15 and 18 of a 28-day course. The dose of ON 01910.Na will be escalated in increments in successive cohorts (dose level (DL) 1 = 600 mg/m2, DL 2 = 1200 mg/m2, DL 3 = 1800 mg/m2) of new patients. A course is defined as 4 weeks in length. Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v3.0). A minimum of three new patients will be treated at each dose level with a minimum of a 1 week stagger between the dosing of the first and remaining patients in each new dose cohort. In exceptional circumstances (e.g. where there is one slot available in a cohort and two eligible patients have been screened), the Sponsor may allow four patients to enter a cohort (or seven patients to enter an expanded cohort). A DL -1A (ON 01910.Na = 400 mg/m2) is set in case dose de-escalation is required with the starting dose due to ON 01910.Na-related toxicity. A DL -1A gemcitabine = 750 mg/m2 and DL - 1B at 500 mg/m2 are set in case dose de-escalation is required with the starting and subsequent doses due to gemcitabine-related toxicity. If DLT is not observed in the first three patients, then the dose of ON 01910.Na will be increased to the next level (see Section 4.2 for definitions of DLT). If DLT occurs in any of the first three new patients in the first course, at least three additional new patients will be treated. If no further DLT is encountered, dose escalation will proceed. Alternately, if DLT is noted in one or more of three additional patients, dose escalation will be terminated and the MTD will be defined as the highest dose level at which none of the first three patients or no more than one of six patients experienced DLT in course 1. All patients receiving doses exceeding the confirmed MTD will have their dose reduced to the MTD; even if apparently tolerating their current dose. Intra-patient dose escalation of ON 01910.Na will be permitted. There will be no limit to the number of courses that could be administered to a patient who is both tolerating and benefiting from therapy.

A patient will be considered evaluable for the purposes of the dose escalation decision if the patient completes the first course of therapy without missing more than 1 dose of ON 01910.Na for reasons unrelated to toxicity, or if the patient is withdrawn due to a DLT. Non-evaluable patients will be replaced. Escalation to the next dose level will occur only after the third evaluable patient (or sixth, if an expanded cohort), on the previous dose level has been observed for 4 weeks. Dose escalation decisions will be made by a Cohort Review Committee (CRC). Intra-patient dose escalation of ON 01910.Na will be allowed after the third evaluable patient on the next dose level has been observed for 4 weeks with acceptable tolerability (ie, MTD has not been exceeded per criteria above).

Once the MTD has been defined, an expanded cohort of 20 to 23 additional patients (depending if 3 or 6 patients were enrolled on the previous cohort) will be enrolled at the MTD dose level in order to further define the safety and tolerability of this regimen, and characterize the pharmacokinetics of ON 01910.Na alone and after gemcitabine, and perform a tumor biomarker study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed solid malignancy for which standard curative or palliative measures do not exist or are no longer effective; or patients with a clinical rationale for a gemcitabine-based therapy.
* The last radiotherapy/chemotherapy dose must have been given ≥4 weeks prior to study drug initiation; with any acute or chronic adverse events of prior radiotherapy or chemotherapy having resolved to <Grade 2 as determined by CTCAE v3.0.
* Patients must have a life expectancy of at least 12 weeks and an ECOG performance status of <1.
* Patients must be >18 years of age.
* Patients must have evaluable disease, either with informative tumor markers, or with measurable disease on imaging, by RECIST (Response Evaluation Criteria in Solid Tumors) criteria (Appendix II).
* Patients must have adequate liver and renal function as defined by serum creatinine no greater than 2.0 times the institution's upper normal limits (or a 24 hour creatinine clearance of >50 ml/min) and total bilirubin level no greater than 2.0 times the institution's upper normal limits and transaminase levels no higher than 3.0 times the institution's upper normal limits. (Note that patients with primary liver cancer or hepatic metastases may have a total bilirubin value of up to 1.5 mg/dl and transaminase levels of up to 5.0 times the limit of normal).
* Patients must have adequate bone marrow function as defined by a granulocyte count of >1,500/mm3, platelet count of >100,000/mm3, and hemoglobin >9 g/dl.
* Patients at the expanded phase at the MTD must be willing and able to undergo blood sampling for pharmacokinetic studies in Course 1.
* For patients in the expanded phase at the MTD, tumor amenable to a single tumor biopsy, and willingness to undergo a baseline tumor biopsy.
* Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study and in keeping with the policies of the institution.

Exclusion Criteria:

Patients will be excluded if:

* They have evidence of active heart disease including myocardial infarction within the previous 3 months; symptomatic coronary insufficiency or heart block; uncontrolled congestive heart failure; moderate or severe pulmonary dysfunction.
* They have an active infectious process.
* They have active central nervous system metastases.
* They have received prior radiotherapy administered to more than 30% of marrow-bearing bone mass.
* They have ascites requiring active medical management including paracentesis more than twice a month or hyponatremia (defined as serum sodium value of <134 Meq/L).
* Women who are pregnant or lactating.
* Male patients with female sexual partners who are unwilling to follow the strict contraception requirements described in this protocol (see Section 5.4).
* Patients who have had major surgery without full recovery or major surgery within 3 weeks of ON 01910.Na treatment start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of treatment to 30 days after end of treatment.
  Incidence of adverse events, including laboratory parameters, as assessed by NCI CTCAE v3.0.
Maximum tolerated dose (MTD) of ON 01910.Na | Escalation phase of protocol.
  MTD will be defined as the highest dose level of ON 01910.Na at which none of the first three patients or no more than one of six patients experienced dose limiting toxicity (DLT) in course 1.

SECONDARY OUTCOMES:
Pharmacokinetics | Confirmation phase of protocol.
  Plasma concentration values of ON 01910.Na will be analyzed to determine if gemcitabine has an effect on pharmacokinetic parameters of ON 01910.Na.
Tumor measurements | Screening to 30 days after end of treatment.
  Tumors will be measured to determine response according to RECIST criteria.
Pharmacodynamics, ex vivo | Confirmation phase of protocol.
  Use tumor tissue obtained by biopsy to assess the pharmacodynamic activity of the ON 01910.Na and gemcitabine combination.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Jimeno, MD, PhD, Study Chair — University of Colorado at Denver Health and Sciences Center
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Denver, Colorado
  - Roswell Park Cancer Institute, Buffalo, New York

REFERENCES:
- [Background] Jimeno A, Li J, Messersmith WA, Laheru D, Rudek MA, Maniar M, Hidalgo M, Baker SD, Donehower RC. Phase I study of ON 01910.Na, a novel modulator of the Polo-like kinase 1 pathway, in adult patients with solid tumors. J Clin Oncol. 2008 Dec 1;26(34):5504-10. doi: 10.1200/JCO.2008.17.9788. Epub 2008 Oct 27. PMID 18955447
- [Background] Jimeno A, Chan A, Cusatis G, Zhang X, Wheelhouse J, Solomon A, Chan F, Zhao M, Cosenza SC, Ramana Reddy MV, Rudek MA, Kulesza P, Donehower RC, Reddy EP, Hidalgo M. Evaluation of the novel mitotic modulator ON 01910.Na in pancreatic cancer and preclinical development of an ex vivo predictive assay. Oncogene. 2009 Jan 29;28(4):610-8. doi: 10.1038/onc.2008.424. Epub 2008 Nov 24. PMID 19029951
- [Background] Jimeno A, Rubio-Viqueira B, Rajeshkumar NV, Chan A, Solomon A, Hidalgo M. A fine-needle aspirate-based vulnerability assay identifies polo-like kinase 1 as a mediator of gemcitabine resistance in pancreatic cancer. Mol Cancer Ther. 2010 Feb;9(2):311-8. doi: 10.1158/1535-7163.MCT-09-0693. Epub 2010 Jan 26. PMID 20103597
- [Result] Ma WW, Messersmith WA, Dy GK, Weekes CD, Whitworth A, Ren C, Maniar M, Wilhelm F, Eckhardt SG, Adjei AA, Jimeno A. Phase I study of Rigosertib, an inhibitor of the phosphatidylinositol 3-kinase and Polo-like kinase 1 pathways, combined with gemcitabine in patients with solid tumors and pancreatic cancer. Clin Cancer Res. 2012 Apr 1;18(7):2048-55. doi: 10.1158/1078-0432.CCR-11-2813. Epub 2012 Feb 14. PMID 22338014
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.